CLINICAL TRIAL: NCT07119723
Title: Environmental Factors and Myopia Prevalence Among Uyghur Students in Remote China
Status: Enrolling by invitation | Type: Observational
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Chuanzhen Zheng, Principal investigator, Tianjin Medical University Eye Hospital
Other Study IDs: 20240902
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Myopia; Environment
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ophthalmologic screening performs annually. Main information collected: gender, age, race, school, visual acuity, autorefractive results.

ELIGIBILITY:
Inclusion Criteria:

* 6 -15 years old

Exclusion Criteria:

* Students with strabismus, amblyopia, or other ocular diseases.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Students aged 6-15 years without strabismus, amblyopia, or other ocular diseases.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent refraction | From January 2020 to December 2026

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hospital, Tianjin, China